CLINICAL TRIAL: NCT04986345
Title: High-intensity Interval Training Prescriptions to Reduce the Risk of Complications Linked to Type 2 Diabetes: the Role of Interval Length on Clinical Benefits and on Physiological Mechanisms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: DT2-HIIT-Prot
Record Dates: First submitted 2021-07-07; First posted 2021-08-02 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes; Ambulatory blood pressure; Continous glucose monitoring; High-intensity interval training; Proteomics; Monocytes; Inflammation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Inflammation | interventions — High-Intensity Interval Training; RE1-silencing transcription factor

STUDY DESIGN:
Intervention Model Description: A semi-randomized (experimental conditions) crossover design will be used with a population of elderly women with T2D, and with three experimental conditions (1- rest, 2-HIIT-10: 10x 1 min, 3- HIIT-4: 4 x 4 min).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rest, HIIT-4, HIIT-10 (Experimental): Both arms start with the rest condition and the order of the two other conditions (HIIT-4 and HIIT-10) is determined at random.
  This arm's sequence of intervention is : 1-Rest; 2- HIIT-4 and 3- HIIT-10.
  Interventions: Other: High-intensity interval training (HIIT)-4; Other: High-intensity interval training (HIIT)-10; Other: Rest
- Rest, HIIT-10, HIIT-4 (Experimental): Both arms start with the rest condition and the order of the two other conditions (HIIT-4 and HIIT-10) is determined at random.
  This arm's sequence of intervention is : 1- Rest; 2- HIIT-10 and 3- HIIT-4.
  Interventions: Other: High-intensity interval training (HIIT)-4; Other: High-intensity interval training (HIIT)-10; Other: Rest

INTERVENTIONS:
Other: High-intensity interval training (HIIT)-4 — 4 intervals of 4 minutes at 90% of maximum cardiac frequency, interspersed with 3-minute rests at 70% of maximum cardiac frequency. The session will last 32 minutes, including warm-up and cooldown.
Other: High-intensity interval training (HIIT)-10 — 10 intervals of 1 minutes at 90% of maximum cardiac frequency, interspersed with 1-minute rests at 70% of maximum cardiac frequency. The session will last 34 minutes, including warm-up and cooldown.
Other: Rest — Participants are to stay seated for 30 minutes while reading or watching television.

SUMMARY:
Type 2 diabetes (T2D) prevalence has steadily been rising in the past decades and its complications, including cardiovascular diseases (CVD), are a major public health concern.

To lower CVD risk and to maintain an adequate glycemic control, Diabetes Canada recommends aerobic exercise of high-intensity interval training (HIIT). The leading hypothesis of this study is that longer intervals will favor an anti-inflammatory immune state, and that and that it will be correlated with reduced arterial stiffness and blood pressure.

DETAILED DESCRIPTION:
Type 2 diabetes (T2D) prevalence has steadily been rising in the past decades and its complications, including cardiovascular diseases (CVD), are a major public health concern. Insulin resistance, an important component of T2D, is associated with vascular dysfunctions, which directly contributes to the pathogenesis of CVD, such as atherosclerosis, and hypertension, particularly with the elderly. It is also suggested that glucose variability, measured with continuous glucose monitors (CGM), is an independent risk factor of CVD in T2D individuals, exposing them to an increased risk of premature death. Moreover, in part because of immune dysregulation, women with T2D are at a heightened risk of developing CVD compared to males. Indeed, monocyte inflammatory profile is altered during the aging process and in women with T2D. This, in turn, causes vascular dysfunction which is associated with a pro-thrombotic state, and exacerbates atherosclerosis and arterial stiffening.

To lower CVD risk and to maintain an adequate glycemic control, Diabetes Canada recommends aerobic exercise of high-intensity interval training (HIIT). However, this recommendation is solely based on the improvement of cardiorespiratory fitness in type 2 diabetes individuals (level of evidence: grade B, level 2). Furthermore, most of these studies use exercise protocols with ergocycles, which limit the ecological validity considering that the elderly population prefers to walk. Though, it is essential to evaluate the impact of different walking HIIT protocols on clinical targets such as arterial pressure, glycemic variability/control using ambulatory blood pressure monitors (ABPM) and CGM.

The preliminary data collected in our laboratory shows that a low volume HIIIT program (6 × 1 min) is insufficient to improve glycemic control/variability and ambulatory blood pressure over 24 hours in elderly diabetic women, despite reducing inflammatory gene expression in monocytes. Interestingly, pro-inflammatory monocytes are linked with hyperglycemia and play a crucial role in the atherosclerotic process, while also being associated with arterial stiffening in individuals with kidney failure, a common T2D complication.

These results raise several questions, including the role played by the length of HIIT intervals on clinical targets. While our preliminary results didn't impact ambulatory blood pressure over 24 hours with shorter intervals (6 × 1 min), other studied showed a reduction of this parameter with longer intervals (4 x 4 min). Therefore, the leading hypothesis of this study is that longer high intensity intervals (Wisløff protocol: 4 x 4 min) will reduce ambulatory blood pressure over 24 hours in a greater extent than shorter intervals (10 x 1 min). Indeed, reduced shear stress induced by shorter intervals could damper cellular and molecular responses to exercise bouts, thereby limiting the effects on arterial stiffness and blood pressure in the hours following exercise. Moreover, changes in gene expression do not guarantee changes at the protein level, and proteins are the real effectors of cellular response. Hence, proteomics will be useful to better understand monocyte response to different HIIT protocols and, possibly, the clinical benefits of this training method. Indeed, longer intervals could induce greater variations to the monocytes' proteome, favoring an anti-inflammatory phenotype, and those changes could be associated with reduced arterial stiffness and blood pressure.

The primary objective of this study is therefore to compare the effect of two treadmill HIIT modalities (4x4 min vs. 10x1 min) on arterial stiffness, ambulatory blood pressure over 24 hours and on glycemic variability in elderly women with T2D. The secondary objective is to assess the proteomic changes in monocytes induced by the two HIIT modalities and to correlate them with changes in clinical parameters.

ELIGIBILITY:
Inclusion Criteria:

* With a diagnostic for type 2 diabetes
* Arterial hypertension (controlled at rest)
* Low or no alcohol consumption (≤ 7 alcoholic beverages/week)
* Non-smoking
* Physically active ( > 60 minutes of structured and scheduled physical activity/week for the previous 3 months)

Exclusion Criteria:

* Insulin therapy
* Use of beta blockers
* Unstable medication in the past 6 months
* Stroke in the past 6 months, or with consequences limiting physical activity practice
* Coronary disease without revascularization, or peripheral artery disease
* Neuropathy, retinopathy of nephropathy diagnostics
* Orthopedic limitations, or medical counter-indication for physical activity practice
* Surgery scheduled during the study period

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-10-04 (Actual); Primary Completion 2023-05-15 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in ambulatory systolic and diastolic blood pressure | During 24 hours after the three experimental conditions (Rest, HIIT-4 and HIIT-10)
  mmHg, measured with an ambulatory blood pressure monitor

SECONDARY OUTCOMES:
Change in arterial stiffness | 30 min post-exercise (in lab measure) and during 24 hours after the three experimental conditions (Rest, HIIT-4 and HIIT-10)
  Estimated using pulse wave velocity (m/s), measured with an ambulatory blood pressure monitor
Change in post-exercise glucose levels | Every 5 min during 2 hours after each experimental condition (Rest, HIIT-4 and HIIT-10)
  Measured with a continuous glucose monitor (mmol/L)
Change in post-prandial glucose levels | during the 2 hour-postprandial time (before and after standardized lunch, as well as at 7.5 , 15, 30 60, 90 and 120 min) for each experimental condition (Rest, HIIT-4, HIIT-10)
  Measured with a continuous glucose monitor and blood samples (mmol/L)
Change in 24h glycemia | During 24 hours after the three experimental conditions (Rest, HIIT-4 and HIIT-10)
  Measured with a continuous glucose monitor (mmol/L)
Change in nocturnal glycemia | During the night, from 10 pm to 7 am following each the three experimental conditions (Rest, HIIT-4 and HIIT-10)
  Measured with a continuous glucose monitor (mmol/L)
Change in time passed in hyperglycemia (> 10 mmol/L) | During 24 hours after each experimental conditions (Rest, HIIT-4 and HIIT-10)
  Measured with a continuous glucose monitor (minutes)
Change in time passed in hypoglycemia (< 3.8 mmol/L) | During 24 hours after each experimental conditions (Rest, HIIT-4 and HIIT-10)
  Measured with a continuous glucose monitor (minutes)
Change in time spent in range (between 3.8 and 10 mmol/L) | During 24 hours after each experimental conditions (Rest, HIIT-4 and HIIT-10)
  Measured with a continuous glucose monitor (minutes)
Change in the proteome of blood monocytes | Before, right after the end and 1hour post exercise (HIIT-4 and HIIT-10)
  Use of proteomics to identify and quantify proteins in isolated peripheral blood monocytes
Change in the proportions of blood monocytes subtypes | Before, right after the end and 1hour post exercise (HIIT-4 and HIIT-10)
  Surface expression of CD14 and CD16, assessed by flow cytometry on isolated monocytes.
Resting systolic and diastolic blood pressure | During the preliminary visit, after 5 min of rest in sitting position
  Measured with a manual sphygmomanometer
Total body weight | At baseline, in fasted state
  Measured with an electric scale (kg)
Height | At baseline, in fasted state
  Measured with an mural stadiometer (m)
Change in monocyte-derived macrophages polarization | Before and right after the end of exercise (HIIT-4 and HIIT-10)
  Surface expression of CD86 and CD206, assessed by flow cytometry on monocyte-derived macrophages differentiated 5 days in vitro.
Change in monocyte-derived macrophages response to lipopolysaccharide (LPS) | Before and right after the end of exercise conditions (HIIT-4 and HIIT-10)
  Monocyte-derived macrophages differentiated 5 days in vitro will be treated or not with LPS for 24h. Culture media will be collected for cytokine secretion determination (Multiplex Luminex)
Change in plasma endothelial nitric oxide synthase (eNOS) | Before, at the end of exercise and 1 hour post-exercise (HIIT-4 and HIIT-10)
  Enzyme-Linked Immunosorbent Assay (ELISA) to quantify the level of human eNOS in plasma (ng/mL).
Change in plasma catecholamines | Before, at the end of exercise and 1 hour post-exercise (HIIT-4 and HIIT-10)
  Enzyme-Linked Immunosorbent Assay (ELISA) to quantify the level of human epinephrine and norepinephrine in plasma (pg/mL).
Change in plasma insulin | during the 2 hour-postprandial time (before and after standardized lunch, as well as at 7.5, 15, 30 60, 90 and 120 min) for each experimental condition (Rest, HIIT-4, HIIT-10)
  Dosage of plasma insulin (pmol/L)
Change in plasma C-peptide | during the 2 hour-postprandial time (before and after standardized lunch, as well as at 7.5, 15, 30 60, 90 and 120 min) for each experimental condition (Rest, HIIT-4, HIIT-10)
  Dosage of plasma C-peptide (ng/mL)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de recherche sur le vieillissement, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ormazabal V, Nair S, Elfeky O, Aguayo C, Salomon C, Zuniga FA. Association between insulin resistance and the development of cardiovascular disease. Cardiovasc Diabetol. 2018 Aug 31;17(1):122. doi: 10.1186/s12933-018-0762-4. PMID 30170598
- [Background] Nalysnyk L, Hernandez-Medina M, Krishnarajah G. Glycaemic variability and complications in patients with diabetes mellitus: evidence from a systematic review of the literature. Diabetes Obes Metab. 2010 Apr;12(4):288-98. doi: 10.1111/j.1463-1326.2009.01160.x. PMID 20380649
- [Background] Shalev V, Chodick G, Heymann AD, Kokia E. Gender differences in healthcare utilization and medical indicators among patients with diabetes. Public Health. 2005 Jan;119(1):45-9. doi: 10.1016/j.puhe.2004.03.004. PMID 15560901
- [Background] Peters SA, Huxley RR, Sattar N, Woodward M. Sex Differences in the Excess Risk of Cardiovascular Diseases Associated with Type 2 Diabetes: Potential Explanations and Clinical Implications. Curr Cardiovasc Risk Rep. 2015;9(7):36. doi: 10.1007/s12170-015-0462-5. PMID 26029318
- [Background] Diabetes Canada Clinical Practice Guidelines Expert Committee; Sigal RJ, Armstrong MJ, Bacon SL, Boule NG, Dasgupta K, Kenny GP, Riddell MC. Physical Activity and Diabetes. Can J Diabetes. 2018 Apr;42 Suppl 1:S54-S63. doi: 10.1016/j.jcjd.2017.10.008. No abstract available. PMID 29650112
- [Background] Amireault S, Baier JM, Spencer JR. Physical Activity Preferences Among Older Adults: A Systematic Review. J Aging Phys Act. 2018 Oct 25:1-12. doi: 10.1123/japa.2017-0234. Online ahead of print. PMID 29283793
- [Background] Shanmugam N, Reddy MA, Guha M, Natarajan R. High glucose-induced expression of proinflammatory cytokine and chemokine genes in monocytic cells. Diabetes. 2003 May;52(5):1256-64. doi: 10.2337/diabetes.52.5.1256. PMID 12716761
- [Background] Roy-Chowdhury E, Brauns N, Helmke A, Nordlohne J, Brasen JH, Schmitz J, Volkmann J, Fleig SV, Kusche-Vihrog K, Haller H, von Vietinghoff S. Human CD16+ monocytes promote a pro-atherosclerotic endothelial cell phenotype via CX3CR1-CX3CL1 interaction. Cardiovasc Res. 2021 May 25;117(6):1510-1522. doi: 10.1093/cvr/cvaa234. PMID 32717023
- [Background] Lee JW, Cho E, Kim MG, Jo SK, Cho WY, Kim HK. Proinflammatory CD14(+)CD16(+) monocytes are associated with vascular stiffness in predialysis patients with chronic kidney disease. Kidney Res Clin Pract. 2013 Dec;32(4):147-52. doi: 10.1016/j.krcp.2013.08.001. Epub 2013 Sep 26. PMID 26877933
- [Background] Ramirez-Jimenez M, Morales-Palomo F, Pallares JG, Mora-Rodriguez R, Ortega JF. Ambulatory blood pressure response to a bout of HIIT in metabolic syndrome patients. Eur J Appl Physiol. 2017 Jul;117(7):1403-1411. doi: 10.1007/s00421-017-3631-z. Epub 2017 May 10. PMID 28493030
- [Background] Ito S. High-intensity interval training for health benefits and care of cardiac diseases - The key to an efficient exercise protocol. World J Cardiol. 2019 Jul 26;11(7):171-188. doi: 10.4330/wjc.v11.i7.171. PMID 31565193
- [Derived] Tremblay R, Marcotte-Chenard A, Deslauriers L, Boulay P, Boisvert FM, Geraldes P, Gayda M, Christou DD, Little JP, Mampuya W, Riesco E. Acute Effect of High-Intensity Interval Exercise on Blood Pressure in Females Living with Type 2 Diabetes and Hypertension. Med Sci Sports Exerc. 2025 May 1;57(5):951-961. doi: 10.1249/MSS.0000000000003639. Epub 2024 Dec 30. PMID 39787496
- [Derived] Low JL, Marcotte-Chenard A, Tremblay R, Islam H, Falkenhain K, Mampuya WM, Mari A, McManus AM, Riesco E, Little JP. An acute bout of 4 x 4-min or 10 x 1-min HIIT improves beta cell glucose sensitivity in postmenopausal females with type 2 diabetes: a secondary analysis. J Appl Physiol (1985). 2025 Jan 1;138(1):311-317. doi: 10.1152/japplphysiol.00777.2024. Epub 2024 Dec 18. PMID 39694495